CLINICAL TRIAL: NCT06341088
Title: Evaluation of Anatomical Results and Sexual Functions After Unilateral and Bilateral Laparoscopic Suture Sacro-hysteropexy Operations, a Prospective Randomised Study
Brief Title: Evaluation of Anatomical Results and Sexual Functions After Unilateral and Bilateral Laparoscopic Suture Sacro-hysteropexy Operations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Gamze Nur Cimilli Şenocak, associate professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/132
Record Dates: First submitted 2024-03-19; First posted 2024-04-02 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Pelvic Organ Prolapse
Keywords: suture sacro hysteropexy; Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- unilateral suture sacro-hysteropexy (Active Comparator): patients in this group will undergo unilateral sacrouterine ligament plication with nonabsorbable suture and unilaterally suspended to the anterior longitudinal ligament.
  Interventions: Procedure: unilateral suture sacro-hysteropexy
- bilateral suture sacro-hysteropexy (Active Comparator): patients in this group will undergo bilateral sacrouterine ligament plication with nonabsorbable sutures and bilaterally suspended to the anterior longitudinal ligament.
  Interventions: Procedure: bilateral suture sacro-hysteropexy

INTERVENTIONS:
Procedure: unilateral suture sacro-hysteropexy — patients in this group will undergo unilateral sacrouterine ligament plication with nonabsorbable suture and unilaterally suspended to the anterior longitudinal ligament.
  Arms: unilateral suture sacro-hysteropexy
Procedure: bilateral suture sacro-hysteropexy — patients in this group will undergo bilateral sacrouterine ligament plication with nonabsorbable suture and bilaterally suspended to the anterior longitudinal ligament.
  Arms: bilateral suture sacro-hysteropexy

SUMMARY:
The study was planned as prospective and randomized. For the study, patients will be randomized into two groups as unilateral and bilateral suture sacro-hysteropexy operations.

DETAILED DESCRIPTION:
The study was planned as prospective and randomized. For the study, patients will be randomized into two groups as unilateral and bilateral suture sacro-hysteropexy operations.Computerized random number table will be used as randomization method. Patients who agree to participate in the study and fulfill the inclusion criteria will be evaluated on the effects of prolapse on quality of life and sexual function before and after the surgical procedures and their complaints and satisfaction will be questioned. Surgical success and complications will be evaluated. Changes in the level of prolapse will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the ages of 18-60
2. No previous prolapse surgery
3. Not having a chronic disease
4. Having stage 3-4 prolapse

Exclusion Criteria:

1. Outside the age range of 18-60 years
2. Previous prolapse surgery
3. Having early stage (1-2) prolapse
4. History of chronic disease

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 64 (Actual)
Dates: Start 2024-04-05 (Actual); Primary Completion 2024-11-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
anatomical success of the operations | changes at 1 and 3 months after surgery
  comparition of preoperative and postoperative pelvic organ prolapse quantification system (POP-Q) measurements of the patients

SECONDARY OUTCOMES:
evaluation of the sexual functions of the patients | changes at 1 and 3 months after surgery
  comparition of preoperative and postoperative FSFI(female sexual function index) scores of the patients

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Nur Cimilli Senocak, Principal Investigator — Ataturk University
Locations (1):
- Atatürk University, Erzurum, Palandöken, Turkey (Türkiye)